CLINICAL TRIAL: NCT06903052
Title: Nurse Parental Support Using a Proactive Mobile App in Symptom Management for Children With Medical Complexity Requiring Mechanical Ventilation: an Effectiveness-implementation Hybrid 2 Study
Brief Title: Nurse Parental Support Using a Proactive Mobile App in Symptom Management for Children With Mechanical Ventilation
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The Hong Kong Polytechnic University (Other)
Responsible Party: Principal Investigator, Dr Winsome Lam, Professor, The Hong Kong Polytechnic University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: SNHongkongPOLYU; Ref: 22231361 (Other Grant/Funding Number: Health and Medical Research Fund)
Record Dates: First submitted 2025-03-14; First posted 2025-03-30 (Actual); Last update posted 2025-06-10 (Actual); Status verified 2025-03

CONDITIONS: Child With Medical Complexity; Symptom Management; Self Efficacy; Mobile Application; Nurse-led Supportive Care
Keywords: parental self-efficacy; children requiring mechanical ventilation; symptom management; mobile application; nurse-led parental support

STUDY DESIGN:
Intervention Model Description: Nurse parental support using a proactive mobile App in symptom management for children requiring mechanical ventilation
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Nurse parental support using a proactive mobile App (Experimental): Nurse parental support using a proactive mobile App in symptom management for children with mechanical ventilation for a 3-month period.
  Interventions: Device: Nurse parental support using a proactive mobile App

INTERVENTIONS:
Device: Nurse parental support using a proactive mobile App — Nurse parental support using a proactive mobile App in symptom management for child with mechanical ventilation

SUMMARY:
The aims of this study are to test the effectiveness of a nurse support using a proactive mobile app to enhance parental self-efficacy in symptom management for children using mechanical ventilations, and alongside identify factors facilitating or deterring the program implementation.

A single group pre-post quasi-experimental study on parents of CMC requiring mechanical ventilation.

Parents will be recruited from a non-government office, with an estimated sample size of 52 parents. Self-administrated questionnaire, and semi-structured interview guide will be used for data collection.

DETAILED DESCRIPTION:
Parents of children required mechanical ventilations at risk of high stress levels because these children have multisystem diseases, including severe neurologic conditions, resulting in potential premature death. Literature suggested that increasing parental self-efficacy in managing their child's symptoms could improve the child's health.

Nurse parental support in symptom management using a proactive mobile health application is an alternative method considered more accessible and nurse-parent interactivity to continue home-based support for the CMC and parents.

Self-administrated questionnaire, and semi-structured interview guide will be used for data collection. Descriptive statistics, including proportions for categorical variables, mean, and SD for normally distributed continuous variables, and median and inter-quartile range for non-normally distributed variables, will be reported. Generalized estimating equation will be used to address the objectives with appropriate link function. Qualitative data will be analyzed using thematic analysis to identify the facilitator, and barriers of program implementation.

ELIGIBILITY:
The inclusion criteria for parents are:

1. parent of a child with mechanical ventilation aged 2-18
2. having a Smartphone
3. able to communicate in Chinese and read Chinese
4. living with his/her child at home.

The exclusion criteria for parents are:

1. a reported mental health disorder
2. engaging in other structured programs related to symptom management 3) living in an area with no internet coverage.

Ages: 2 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 52 (Estimated)
Dates: Start 2025-05-06 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2028-04-30 (Estimated)

PRIMARY OUTCOMES:
Caregiving Self-efficacy | Day 0, Month 3, Month 6, Month 9
  The scale consists of 18 items to measure the self-efficacy of Chinese caregivers. It is rated on a 9-point scale, with 1= no confidence, to 9 =full confidence.
Implementation evaluation | month 9
  Semi-structured interviews will be conducted to the related community stakeholders to evaluate the quality of service provided. Semi-structured interview guide will be used to collect qualitative data in four perspectives including:
  1. reach: document the number of participants, and retention in the intervention
  2. adoption: seek to find out if the intervention is appropriate and in action
  3. implementation: understand stakeholders' perception if the intervention is acceptable and implemented as planned
  4. maintenance: explore the facilitators and barriers in the sustainability of the nurse parental support using a proactive mobile app

SECONDARY OUTCOMES:
Modified Memorial Symptom Assessment Scale | Day 0, Month 3, Month 6, Month 9
  This is a modified 40-item Memorial Symptom Assessment Scale (MSAS in Chinese version). The items for measuring the frequency and severity of symptoms are rated on a 4-point Likert scale from one (almost never) to four (always). The items for measuring distress are rated on a 5-point Likert scale from one (not at all) to five (very).
Children health service utilization | Day 0, Month 3, Month 6, Month 9
  This is a record used to summarize a child's visits to outpatient clinic and emergency room, and the child's admission history.

CONTACTS AND LOCATIONS:
Overall Officials: Winsome LAM, PhD, Principal Investigator — The Hong Kong Polytechnic University
Locations (1):
- School of Nursing The Hong Kong Polytechnic University, Kowloon, Kowloon, Hong Kong

IPD SHARING:
Plan to Share IPD: No
IPD collected throughout the study, only IPD used in the results publication